CLINICAL TRIAL: NCT02481115
Title: Pediatric Delirium in Infants and Young Children: Validation of the PreSchool Confusion Assessment Method for the Intensive Care Unit (psCAM-ICU)
Brief Title: Validation of the PreSchool Confusion Assessment Method for the Intensive Care Unit (psCAM-ICU)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Heidi A. Beverley Smith, Assistant Professor of Anesthesiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 121252
Record Dates: First submitted 2015-06-18; First posted 2015-06-25 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Delirium; Cognitive Impairment
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically Ill Children: Children in the Pediatric Critical Care Unit regardless of admitting diagnosis aged at least 6 months of age up to 5 years of age.

SUMMARY:
The investigators hypothesize that critical care trained registered nurses and physicians can perform measurements of cognitive impairment in critically ill pediatric patients in a reliable and valid manner. To test this hypothesis, the investigators will incorporate an instrument (psCAM-ICU) to assess both components of consciousness, arousal and content, in critically ill pediatric patients at least 6 months to children 5 years of age, both on and off mechanical ventilation, and compare these assessments to those of the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Pediatric Critical Care Unit regardless of admitting diagnosis aged at least 6 months of age up to 5 years of age.
* Patients ventilated or non-ventilated.

Exclusion Criteria:

* Non-English speaking patients.
* Children with visual or hearing impairments.
* Patient/surrogate or physician refusal
* Moribund and not expected to survive >48 hours
* Patients in whom comfort care orders have been instituted
* Patients who are identified for transfer to floor or home regardless of placed orders or bed availability

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically ill pediatric patients at least 6 months to children 5 years of age, both on and off mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Validation of psCAM-ICU | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The investigators will validate the psCAM-ICU against a reference standard delirium assessment in critically ill infants and young children. Critical care physicians and registered nurses will use the psCAM-ICU to determine presence or absence of delirium once daily in critically ill infants and young children from 6 months to less than 5 years of age. The reference standard, a pediatric delirium expert (child psychiatrist or equivalent), will independently evaluate the same patients for presence or absence of delirium using the Diagnostic and Statistical Manual of Mental Disorders (DSM IV-TR) as the foundation of assessment.

SECONDARY OUTCOMES:
Inter-rater reliability of diagnosing delirium | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The investigators will assess inter-rater reliability between physician, practitioner, and nursing assessment using the psCAM-ICU. The psCAM-ICU should consistently diagnose delirium in the critically ill pediatric patient, independent of the type of medical care provider assessing the patient.
Validation of the Richmond Agitation Sedation Scale (RASS) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The investigators will validate the RASS against the Glasgow Coma Scale in critically ill infants and young children less than 5 years of age.
Validation of the Withdrawal Assessment Tool-1 (WAT-1) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The investigators will validate the WAT-1 against a reference standard (child psychiatrist) in critically ill infants and young children less than 5 years of age.
Long-term cognitive impairment composite | 1 year
  Clinical data will be obtained from the medical record to determine a composite measure of long-term cognitive impairment. The composite will include specific outcomes, and follow-up phone interviews with be conducted with a parent/legal guardian at 12 months post-hospital discharge of enrolled patients to assess cognitive function using a validated questionnaire that is compared to expected developmental trajectories based on age adjusted norms.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Smith, MD, Principal Investigator — Vanderbilt University School of Medicine

IPD SHARING:
Plan to Share IPD: No